CLINICAL TRIAL: NCT05399849
Title: Acceptability, Feasibility, Usability, and Effectiveness of a Mindfulness Intervention in Young Adults With a Concussion History: A Pilot Study
Brief Title: Mindfulness Intervention in Young Adults With a Concussion History
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0732
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-08

CONDITIONS: Concussion, Brain; Concussion Post Syndrome
Keywords: Concussion; Mindfulness; Intervention; Perceived Stress
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome | interventions — Meditation

STUDY DESIGN:
Masking Description: This pilot study has no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Intervention (Experimental): All participants will be enrolled in the mindfulness intervention arm to complete the six-week mindfulness intervention.
  Interventions: Behavioral: Mindfulness Exercises and Meditations

INTERVENTIONS:
Behavioral: Mindfulness Exercises and Meditations — Mindfulness exercises will be completed independently using the LoveYourBrain Foundation Meditation Library, a free, online resource containing traumatic brain injury-focused mindfulness-focused exercises and meditations. Mindfulness-based exercises and meditations to be completed will be chosen by study personnel based on tools utilized in mindfulness-based stress reduction programs that are provided on the LoveYourBrain Meditation Library. Specific mindfulness-based exercises and meditations will include body scan, acceptance, awareness, and breathing.

SUMMARY:
Young adults (aged 18-30) with a concussion history (defined as experiencing a concussion within the past five years but not within the past month) will complete a six-week mindfulness intervention. Throughout the intervention, participants will complete 10-20 minutes of mindfulness-focused exercises and meditations each day using the LoveYourBrain Foundation Meditation Library. Before the intervention, participants will complete a baseline assessment including demographics, concussion history, mental health history, mindfulness history, perceived stress, mindfulness, and concussion symptoms. Throughout the intervention, participants will complete weekly assessments measuring adherence and concussion symptoms. After six weeks, participants will complete a final, follow-up assessment with assessments for adherence, acceptability, feasibility, intervention perceptions, perceived stress, mindfulness, and concussion symptoms.

This study's aim is to determine the acceptability, feasibility, usability, and effectiveness of a mindfulness intervention in young adults with a concussion history. The investigators hypothesize that participants who participate in the mindfulness intervention will report high adherence (complete five days of meditation per week), positive acceptability, positive feasibility, and positive intervention perceptions. Additionally, after completing the intervention, participants will report decreased perceived stress, increased mindfulness, and decreased concussion symptoms compared to before the intervention.

DETAILED DESCRIPTION:
This study is a pilot prospective, feasibility intervention clinical trial. As this is a novel, pilot intervention in the proposed population, the study will utilize an uncontrolled study design where all participants will partake in the six-week, longitudinal mindfulness intervention. All participants will be recruited via the University of North Carolina at Chapel Hill and all data will be collected via the single site. Participants will complete baseline measures for concussion symptoms, perceived stress, and mindfulness. For the six-week intervention, participants will complete 10-20 minutes of mindfulness-focused exercises and meditations each day. Mindfulness exercises will be completed independently using the LoveYourBrain Foundation Meditation Library, a free, online resource containing traumatic brain injury-focused mindfulness-focused exercises and meditations. Mindfulness-based exercises and meditations to be completed will be chosen by study personnel based on tools utilized in mindfulness-based stress reduction programs that are provided on the LoveYourBrain Meditation Library. Specific mindfulness-based exercises and meditations will include body scan, acceptance, awareness, and breathing. At intervention enrollment participants will be presented with a detailed manual providing them with beginner mindfulness tips and instructions as well as details on the purpose for the intervention. Before beginning the exercises and after being presented the manual, participants will be asked by study personnel if they have any questions or concerns regarding the intervention. Throughout the six-week intervention, study personnel will prompt participants via email and text at the beginning of each week with the specific exercises/meditations to be completed each day for that week. Participants will be prompted via email and text at the end of each week to complete a questionnaire to assess adherence and track concussion symptoms. Participants will have one day to complete the weekly assessment. If it is not completed on that day, study personnel will prompt the participant via email and text for three days. If the assessment is not completed in three days, study personnel will call participants to complete the assessment. At three weeks (halfway through the intervention), study personnel will call participants to complete the weekly assessment and check in on participation. Upon completion of the six-week trial, participants will be prompted via email and text to complete a final assessment including questions regarding adherence, acceptability, feasibility, intervention perceptions, concussion symptoms, perceived stress, and mindfulness. Participants will have one day to complete the final assessment. If they have not completed the final assessment at that time, study personnel will prompt the participant via email and text for three days. If it is not completed after three days, study personnel will call the participant to complete the assessment over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18-30
* Concussion history (defined as experiencing a concussive injury within the past five years, but not within the past month)

Exclusion Criteria:

* History of moderate and/or severe traumatic brain injury
* Currently under provider care for a concussion/traumatic brain injury
* Health risks (heart conditions, respiratory disorders, and/or neurological disorders) that put them at greater than minimal risk
* Current mindfulness practice
* There will be no exclusion based on self-report sex, race, ethnicity, or mental health history.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Mean Acceptability of Intervention (AIM) Total Score | Follow-up (post-intervention, week 6) approximately 42 days after intervention initiation.
  Acceptability will be assessed during the post-intervention follow-up (week 6) assessment using the AIM. The AIM is a four-item validated measure assessing associations with an intervention. It is assessed on a five-point scale from 1=completely disagree to 5=completely agree. A total score will be computed by summing the responses for all four items (higher scores indicating more positive acceptance). The outcome for acceptability will be the AIM total score (range=4-20). The mean AIM total score for all participants will be reported.
Mean Feasibility of Intervention (FIM) Total Score | Follow-up (post-intervention, week 6) approximately 42 days after intervention initiation.
  Feasibility will be measured during the post-intervention follow-up (week 6) assessment using the FIM, a four-item validated measure assessing intervention feasibility. The FIM is assessed on a five-point scale from 1=completely disagree to 5=completely agree. A total score will be computed by summing the responses for all four items (higher scores indicating more positive feasibility). The outcome for feasibility will be the FIM total score (range=4-20). The mean FIM total score for all participants will be reported.

SECONDARY OUTCOMES:
Mean Days of Mindfulness Exercises/Meditations Completed Per Week | Approximately 7 to 42 days after intervention initiation.
  Throughout the intervention participants will be prompted to complete a weekly questionnaire to assess adherence. Subjects will be asked which mindfulness exercises/meditations they completed for that week. Adherence will be assessed at weeks 1, 2, 3, 4, 5, and 6 (post-intervention follow-up). The outcome for adherence will be the number of days of mindfulness exercises/meditations completed per week (range=0-7). The mean number of days of mindfulness exercises/meditations completed per week for all participants will be reported.
Mean Rivermead Post-Concussion Questionnaire (RPQ) Symptom and Severity Score | Baseline (pre-intervention, week 0).
  Concussion symptoms will be measured using the RPQ, a validated measure which asks participants to report the presence and severity (0-4) of 18 concussion-related symptoms compared with before their concussion. The RPQ has been frequently used in the study population. Concussion symptoms will be assessed at baseline (pre-intervention, week 0) and follow-up (post-intervention, week 6). Outcomes for concussion symptoms will include the total symptoms (range=0-18) and total symptom severity (range=0-72) reported from the RPQ. The mean RPQ total symptoms and total symptom severity for all participants will be reported.
Mean Rivermead Post-Concussion Questionnaire (RPQ) Symptom and Severity Score | Follow-up (post-intervention, week 6). Approximately 42 days after intervention initiation.
  Concussion symptoms will be measured using the RPQ, a validated measure which asks participants to report the presence and severity (0-4) of 18 concussion-related symptoms compared with before their concussion. The RPQ has been frequently used in the study population. Concussion symptoms will be assessed at baseline (pre-intervention, week 0) and follow-up (post-intervention, week 6). Outcomes for concussion symptoms will include the total symptoms (range=0-18) and total symptom severity (range=0-72) reported from the RPQ. The mean RPQ total symptoms and total symptom severity for all participants will be reported.
Mean Perceived Stress Scale (PSS-10) Total Score | Baseline (pre-intervention, week 0).
  Perceived stress will be measured using the PSS-10, the most widely used psychological instrument for measuring perceived stress. The PSS-10 is well validated and had been used in connection to mindfulness and in brain injury populations. The PSS-10 consists of 10 questions on a five-point scale (0=never to 4=very often) about how often a participant has felt or thought a certain way relative to their perceived stress in the past month. Final scores will be obtained by reversing responses to the four positively stated items and then summing all 10 scale items (higher scores indicate higher perceived stress). Perceived stress will be assessed at baseline (pre-intervention, week 0) and follow-up (post-intervention, week 6). The outcome for perceived stress will be the PSS-10 total score (range=0-40). The mean PSS-10 total score for all participants will be reported.
Mean Perceived Stress Scale (PSS-10) Total Score | Follow-up (post-intervention, week 6). Approximately 42 days after intervention initiation.
  Perceived stress will be measured using the PSS-10, the most widely used psychological instrument for measuring perceived stress. The PSS-10 is well validated and had been used in connection to mindfulness and in brain injury populations. The PSS-10 consists of 10 questions on a five-point scale (0=never to 4=very often) about how often a participant has felt or thought a certain way relative to their perceived stress in the past month. Final scores will be obtained by reversing responses to the four positively stated items and then summing all 10 scale items (higher scores indicate higher perceived stress). Perceived stress will be assessed at baseline (pre-intervention, week 0) and follow-up (post-intervention, week 6). The outcome for perceived stress will be the PSS-10 total score (range=0-40). The mean PSS-10 total score for all participants will be reported.
Mean Five Facet Mindfulness Questionnaire (FFMQ) Total Score | Baseline (pre-intervention, week 0).
  Mindfulness will be measured using the FFMQ. This widely used, valid survey to measure mindfulness has been researched extensively connected to perceived stress. Participants will be asked 39 questions on a five-point scale (1=never/very rarely true to 5=very often/always true) related to general mindfulness tendencies in daily life. Final scores will be obtained by reversing responses to the 19 reverse scored questions and then summing all 39 items (higher scores indicate greater mindfulness levels). Mindfulness will be assessed at baseline (pre-intervention, week 0) and follow-up (post-intervention, week 6). The outcome for mindfulness will be the FFMQ total score (range=39-195). The mean FFMQ total score for all participants will be reported.
Mean Five Facet Mindfulness Questionnaire (FFMQ) Total Score | Follow-up (post-intervention, week 6). Approximately 42 days after intervention initiation.
  Mindfulness will be measured using the FFMQ. This widely used, valid survey to measure mindfulness has been researched extensively connected to perceived stress. Participants will be asked 39 questions on a five-point scale (1=never/very rarely true to 5=very often/always true) related to general mindfulness tendencies in daily life. Final scores will be obtained by reversing responses to the 19 reverse scored questions and then summing all 39 items (higher scores indicate greater mindfulness levels). Mindfulness will be assessed at baseline (pre-intervention, week 0) and follow-up (post-intervention, week 6). The outcome for mindfulness will be the FFMQ total score (range=39-195). The mean FFMQ total score for all participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Callahan, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Approval from an IRB, IEC or REB and an executed data use/sharing agreement with the UNC-Chapel Hill.